CLINICAL TRIAL: NCT04992052
Title: A Prospective, Randomized, Single-blinded Superiority Study to Evaluate Bone Wax Use for Hemostasis During Primary Unilateral Total Knee Arthroplasty
Brief Title: Bone Wax Use for Hemostasis During Primary Unilateral Total Knee Arthroplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor Enrollment
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Eugene Krauss, Director of Orthopaedics, Syosset Hospital, Northwell Health System, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-0044-NSUH
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Results first posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Total Knee Replacement
Keywords: Knee arthroplasty; Total knee replacement

STUDY DESIGN:
Intervention Model Description: Arm 1 Bone wax applied to the exposed cancellous surfaces of the bone (treatment group).
  Arm 2 No bone wax. This group will serve as the control arm.
Who Masked: Participant, Care Provider
Masking Description: Blinding of the principal investigator and operating staff is not possible. However, all attempts will be made to keep this information from the hospital staff caring for the patients in the postoperative period. The patient and the postoperative hospital staff will be blinded to the treatment arm. The OR staff will be trained not to discuss this information with the patient. During the transition of care from the OR to the Post Anesthetic Care Unit (PACU) the treatment arm will not be included in the verbal patient report. The lack of this information is not required to effectively manage the patient in the postoperative period and will not affect patient care. Postoperatively medical care is managed by the hospitalist, medical doctors specializing in the care of hospitalized patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment arm (Active Comparator): This arm will have bone wax applied to the exposed cancellous surfaces of the bone.
  Interventions: Device: Bone wax
- Control Arm (No Intervention): This arm will serve as the control group. Bone wax will not be used in this group.

INTERVENTIONS:
Device: Bone wax — The surgeons will apply the bone wax to the exposed cancellous bone after the implant has been cemented in place in patients randomized to the treatment arm.
  Arms: Treatment arm

SUMMARY:
The purpose of this study is to assess whether the application of bone wax to exposed cancellous bone, after the cemented implants are in place, will provide superior hemostasis in total knee arthroplasty (TKA) patients compared to patients who do not have the bone wax applied. Hemostasis will be assessed by calculating blood loss using the Hb-balance formula.

DETAILED DESCRIPTION:
Total joint arthroplasty can result in significant blood loss. Postoperative anemia has been associated with prolonged length of stay and increased hospital costs.1 Minimizing blood loss has led to multiple blood conservation strategies in orthopaedic procedures.

Bone wax is a well-known topical hemostatic agent comprised of a mixture of beeswax, paraffin, and isopropyl palmitate. This inexpensive agent works by sealing the bleeding site and tamponades bleeding from the cancellous bone. Bone wax can be precisely applied evenly and stops bone bleeding immediately upon application.2

The purpose of this study is to assess whether the application of bone wax to exposed cancellous bone, after the cemented implants are in place, will provide superior hemostasis in total knee arthroplasty (TKA) patients compared to patients who do not have the bone wax applied. Hemostasis will be assessed by calculating blood loss using the Hb-balance formula.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for primary unilateral total knee arthroplasty
2. Preoperative Hemoglobin >11mg/dL
3. Preoperative platelet count of >150,000

Exclusion Criteria:

1. Patients unable to take aspirin or apixaban for VTE prophylaxis
2. Allergy to any of the ingredients in bone wax (beeswax, paraffin, or isopropyl palmitate)
3. Patients taking clopidogrel (Plavix), ticagrelor (Brilinta), or prasugrel (Effient) or any other antiplatelet medication (except for aspirin 81 mg)
4. Patients unable to get IV Tranexamic Acid for any reason
5. Patients requiring anticoagulant treatment prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Krauss, MD, Principal Investigator — Syosset Hospital, Northwell Health
Locations (1):
- Syosset Hospital, Syosset, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shin KH, Choe JH, Jang KM, Han SB. Use of bone wax reduces blood loss and transfusion rates after total knee arthroplasty. Knee. 2020 Oct;27(5):1411-1417. doi: 10.1016/j.knee.2020.07.074. Epub 2020 Aug 19. PMID 33010755
- [Background] Noble PC, Scuderi GR, Brekke AC, Sikorskii A, Benjamin JB, Lonner JH, Chadha P, Daylamani DA, Scott WN, Bourne RB. Development of a new Knee Society scoring system. Clin Orthop Relat Res. 2012 Jan;470(1):20-32. doi: 10.1007/s11999-011-2152-z. PMID 22065240
- [Result] Moo IH, Chen JYQ, Pagkaliwaga EH, Tan SW, Poon KB. Bone Wax Is Effective in Reducing Blood Loss After Total Knee Arthroplasty. J Arthroplasty. 2017 May;32(5):1483-1487. doi: 10.1016/j.arth.2016.12.028. Epub 2016 Dec 24. PMID 28089184

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was terminated early due to slow enrollment.
Period: Overall Study
Arm/Group | Treatment Arm | Control Arm
Started | 29 | 23
Completed | 29 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm | Control Arm | Total
Number analyzed (Participants) | 29 | 23 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 14 | 8 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 17 | 38
  Male | 8 | 6 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Blood Loss
Description: To determine if there is a change in blood volume loss between the two study arms.
Time Frame: Blood loss is measured the morning of postoperative day 1.
Population: One patient in the control arm did not have any blood work done on postoperative day 1, therefore, the blood loss analysis could not be calculated.
Measure: Mean (Standard Deviation); unit: mililiters
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 29 | 22
mililiters | 810.48 (342.47) | 905.36 (371.92)

2. Secondary Outcome: Knee Society Scoring System
Description: To determine if there is a change in patient functional outcomes, as measured by the Knee Society Scoring System, between the two study arms. The minimum and maximum score for this scale ranges from 0-100. A higher score means a better outcome.
Time Frame: The Knee Society Score was collected within two months prior to the day of surgery and on postoperative day 56 with a collection window of +/- 2 weeks.
Population: 7 patients in the treatment arm and 4 patients in the control arm did not complete the postoperative knee society score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 22 | 19
score on a scale | 62.55 (19.42) | 56.32 (15.36)

ADVERSE EVENTS:
Time Frame: Patients were followed for 90 days after the day of surgery for any adverse events or device related events.
Arm/Group | Treatment Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/23
Other Adverse Events (participants affected / at risk) | 0/29 | 0/23

LIMITATIONS AND CAVEATS:
This study was terminated early due to poor enrollment. In order to do formal power calculation using a two-sample t-test at a significance level of 0.05, a sample size of 100 subjects would be needed to detect a difference in mean blood loss of about 150 mL to 200 mL between the control group and the treatment group. A blood loss of 150 mL to 200 mL is the value which the investigators consider to be clinically significant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/52/NCT04992052/Prot_SAP_000.pdf